CLINICAL TRIAL: NCT03415035
Title: Venetoclax in Chronic Lymphocytic Leukemia Effectiveness and Real-life Treatment Management
Brief Title: Study Venetoclax Effectiveness and Real-Life Treatment Management in Participants With Chronic Lymphocytic Leukemia
Acronym: VERONE
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-913
Record Dates: First submitted 2018-01-24; First posted 2018-01-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cancer - Chronic Lymphocytic Leukemia
Keywords: Venetoclax; Venclyxto; Cancer; Chronic Lynmphocytic Leukemia (CLL)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Chronic Lymphocytic Leukemia (CLL): Patients with diagnosed CLL and eligible to venetoclax as per label

SUMMARY:
This study will evaluate real-life effectiveness and use in participants starting venetoclax treatment for Chronic Lymphocytic Leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosed Chronic Lymphocytic Leukemia (CLL) and eligible for venetoclax as per label.
* Participants for whom the physician has decided to initiate CLL treatment with venetoclax.
* Participants the physician believes he can personally follow over all the study period.
* Participants who have been informed verbally and in writing about this study, and who do not object to their data being electronically processed or subjected to data quality control.

Exclusion Criteria:

- Participating in a clinical trial with an investigative drug for CLL within 30 days prior to treatment initiation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients starting venetoclax treatment for CLL.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Best Response of Venetoclax in Participants with Chronic Lymphocytic Leukemia (CLL) up to 12 Months | Up to approximately 12 months
  The best response is defined as the best response observed during the first year of study treatment among the possible responses to treatment: Complete Response (CR), CR with incomplete bone marrow recovery (CRi), nodular Partial Response (nPR), Partial Response (PR), Stable Disease (SD), or Disease Progression (DP).

SECONDARY OUTCOMES:
Time To Next Treatment | Up to approximately 48 months
  The time to next treatment is defined as the time between the date of the first venetoclax intake and the date of the first next treatment intake after venetoclax discontinuation.
Time to First Response to Treatment (TTR) | Up to approximately 24 months
  The time to response to treatment (TTR) is defined by the time between the date of the first venetoclax intake and the date of the first assessment having documented the response among CR, CRi, nPR, and PR.
Minimal Residual Disease | Up to approximately 24 months
  The proportion of participants with assessment of the minimal residual disease under venetoclax treatment (assessed by flow cytometry or Polymerase Chain Reaction).
Overall Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the proportion of participants who reach either CR, CRi, nPR, or PR to treatment, according to physician's assessment.
Change in Score of EuroQol 5 Dimensions (EQ-5D-5L) | Up to approximately 24 months
  The EQ-5D-5L has five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. These dimensions are measured on a five-level scale: no problems, slight problems, moderate problems, severe problems, and extreme problems. The scores for the 5 dimensions are used to compute a single utility index score ranging from zero (0.0) to 1 (1.0) representing the general health status of the individual. The EQ-5D-5L also contains a visual analog scale (VAS) to assess the subject's overall health.
Time to Best Response to Treatment | Up to approximately 24 months
  The time to best response to treatment is defined by the time between the date of the first venetoclax intake and the date of the assessment having documented the best response among CR, CRi, nPR, PR, SD, and DP.
Response Duration | Up to approximately 48 months
  The response duration will be calculated in the sub-population of participants experiencing treatment response (CR, CRi, nPR, or PR) from the date when response is first met to the date of first following documented progression.
PFS after Disease Progression Following Venetoclax Treatment | Up to approximately 48 months
  The PFS after disease progression following venetoclax treatment will be calculated in the sub-population of patients experiencing disease progression under venetoclax. The PFS following venetoclax treatment is defined as the time from the date of first next CLL treatment intake to the date of the following documented progression or death from any cause.
Overall survival (OS) | Up to approximately 48 months
  OS is defined as the time from the date of first venetoclax intake to the date of death from any cause.
Best Response under Next CLL Treatment | Up to approximately 48 months
  The best response under next CLL treatment will be calculated in the sub-population of patients having a next CLL treatment after venetoclax discontinuation.
Progression-Free Survival (PFS) | Up to approximately 48 months
  PFS is defined as the time from the date of first venetoclax intake to the date of the first documented disease progression or death from any cause.
Time To Progression (TTP) | Up to approximately 48 months
  The Time To Progression (TTP) is defined as the time from the date of first venetoclax intake to the date of the first documented disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (60):
- France (60):
  - CH Cannes - les Broussailles /ID# 201108, Cannes, Alpes-Maritimes
  - CH CARCASSONNE - Antoine Gayraud /ID# 202530, Carcassonne, Aude
  - CHU Clermont-Ferrand /ID# 170736, Clermont, Auvergne-Rhône-Alpes
  - Clinique Pole santé République /ID# 204658, Clermont-Ferrand, Auvergne
  - CH de la Haute-Saône - Vesoul /ID# 205150, Vesoul, Bourgogne-Franche-Comté
  - CHU de RENNES /ID# 169944, Rennes, Brittany Region
  - CHU de Besancon - Jean Minjoz /ID# 170721, Besançon, Doubs
  - Centre Hospitalier de Cornouaille /ID# 169937, Quimper, Finistere
  - CHU Limoges - Dupuytren 1 /ID# 200193, Limoges, Franche-Comte
  - Institut Bergonie /ID# 170746, Bordeaux, Gironde
  - CH Roubaix - Hopital Victor Provo /ID# 170909, Roubaix, Hauts-de-France
  - CHU Montpellier - Hopital Saint Eloi /ID# 200192, Montpellier, Herault
  - CH de Saint-Malo - Hôpital Broussais /ID# 169935, St-Malo, Ille-et-Vilaine
  - CHRU Tours - Hopital Bretonneau /ID# 169469, Tours, Indre-et-Loire
  - CHU Grenoble - Hopital Michallon /ID# 170741, La Tronche, Isere
  - CHU Reims - Hôpital Robert Debre /ID# 170917, Reims, Marne
  - CHRU Nancy - Hopitaux de Brabois /ID# 170855, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CH Bretagne Atlantique /ID# 200191, Vannes, Morbihan
  - CHR Metz-Thionville - Hopital Bel-Air /ID# 170722, Thionville, Moselle
  - IUCT Oncopole /ID# 170749, Toulouse, Occitanie
  - AP-HP - Hopital Bicetre /ID# 170747, Le Kremlin-Bicêtre, Paris
  - Hopital de la Conception /ID# 201981, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de la Cote Basque /ID# 170735, Bayonne, Pyrenees-Atlantiques
  - Centre Leon Berard /ID# 170018, Lyon, Rhone
  - Clinique Victor Hugo /ID# 169973, Le Mans, Sarthe
  - Centre Hospitalier du Mans /ID# 169451, Le Mans, Sarthe
  - Hopital de Melun /ID# 202569, Melun, Seine-et-Marne
  - Centre Henri Becquerel /ID# 169948, Rouen, Seine-Maritime
  - CHU Amiens-Picardie Site Sud /ID# 170724, Amiens, Somme
  - Institut Gustave Roussy /ID# 202436, Villejuif, Val-de-Marne
  - CHU Poitiers - La miletrie /ID# 169470, Poitiers, Vienne
  - CHI POISSY - Saint-Germain-en-Laye /ID# 169966, Saint-Germain-en-Laye, Yvelines
  - Ch Agen /Id# 170742, Agen
  - CH Victor Dupouy /ID# 169946, Argenteuil
  - Ch Blois /Id# 170727, Blois
  - CHRU de Brest - Hopital Morvan /ID# 169457, Brest
  - CHU de CAEN - Hopital de la Cote de Nacre /ID# 169941, Caen
  - Hopital Prive Sevigne /Id# 170718, Cesson-Sévigné
  - Medipole de Savoie /ID# 169454, Challes-les-Eaux
  - CH William Morey /ID# 169939, Chalon-sur-Saône
  - Centre Hospitalier de CHOLET /ID# 171215, Cholet
  - Hopital d'Instruction des Armées PERCY /ID# 170740, Clamart
  - Centre Joseph BELOT /ID# 170853, Désertines
  - CH Annecy Genevois - Site Annecy /ID# 200826, Epagny Metz Tessy
  - Centre Hospitalier de Versailles André Mignot /ID# 169950, Le Chesnay
  - CH Libourne - Hopital Robert Boulin /ID# 170739, Libourne
  - Hopital Saint Vincent de Paul /ID# 169956, Lille
  - Clinique de la Sauvegarde /ID# 169904, Lyon
  - CH Princesse Grace /ID# 200196, Monaco
  - CH Mont de MARSAN /ID# 169955, Mont-de-Marsan
  - Ch Mulhouse /Id# 170726, Mulhouse
  - Polyclinique le LANGUEDOC /ID# 169925, Narbonne
  - Centre Hospitalier Régional d'Orléans - Hôpital de la Source /ID# 169453, Orléans
  - Hôpital Saint-Louis /ID# 170856, Paris
  - Centre Hospitalier de Perpignan /ID# 170743, Perpignan
  - CH Périgueux /ID# 169458, Périgueux
  - CH Saint-Brieuc /ID# 171076, Saint-Brieuc
  - Hopital Nord Franche Comté /ID# 170744, Trévenans
  - Hopital Avicenne - APHP /ID# 169940, Bobigny, Île-de-France Region
  - Hopital Pitie Salpetriere /ID# 169974, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com/